CLINICAL TRIAL: NCT04053010
Title: A Randomized, Controlled, Multicenter Vaccine Clinical Trial to Evaluate The Safety and Immunogenicity of Combined Immunization With sIPV and DTaP
Brief Title: Clinic Trial to Evaluate the Safety and Immunogenicity of Combined Immunization of sIPV and DTaP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Wuhan Institute of Biological Products Co., Ltd (Industry); Beijing Institute of Biological Products Co Ltd. (Industry); Shaanxi Provincial Center for Disease Control and Prevention (Other); Hubei Provincial Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: sIPV/DTaP-2019-02
Record Dates: First submitted 2019-08-09; First posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Vaccination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1 (Experimental): 234 subjects; simultaneously administration of Sabin-IPV and DTaP at the age of 3/4/5 months old, 0.5 ml each dose, respectively
  Interventions: Biological: Sabin-IPV and DTaP
- group 2 (Active Comparator): 234 subjects; Sabin-IPV only at the age of 3/4/5 months old, 0.5 ml each dose, respectively
  Interventions: Biological: Sabin-IPV
- group 3 (Active Comparator): 234 subjects; DTaP only at the age of 3/4/5 months old, 0.5 ml each dose, respectively
  Interventions: Biological: DTaP

INTERVENTIONS:
Biological: Sabin-IPV and DTaP — Sabin-IPV +DTaP at the age of 3/4/5 months old respectively
  Arms: group 1
Biological: Sabin-IPV — Sabin-IPV only at the age of 3/4/5 months old respectively
  Arms: group 2
Biological: DTaP — DTaP only at the age of 3/4/5 months old respectively
  Arms: group 3

SUMMARY:
Eligible,healthy infants will be recruited and divided into 3 groups:(1)combined immunization of sIPV and DTaP group, (2) sIPV group and (3) DTaP group. After completing the two basic vaccine EPI procedures, the immunogenicity and safety of the combined immunization group and the individual vaccination groups will be compared and analyzed.

DETAILED DESCRIPTION:
It is recommended by China Food and Drug Administration (CFDA) that studies on simultaneous immunization of Sabin-IPV and DTaP be carried out as soon as possible, and the immunogenicity and safety studies should also be conducted. Currently in China the vaccination schedules of sIPV and DTaP overlap at infants' 3rd and 4th months of age. In order to avoid the vaccination time conflict and explore the possibility of simultaneous vaccination, we design this clinical study of simultaneous vaccination of the two vaccines.

To be specific, the subjects were divided into 3 groups. Group 1 : sIPV (1st, 2nd, and 3rd doses) and DTaP (1st, 2nd, and 3rd doses) were simultaneously inoculated at 3,4,5 months old ; Group 2 : received 1 dose of sIPV at 3,4,5 months old ; Group 3 : received 1 dose of DTaP at 3,4,5 months old . Blood sample would be collected both before vaccination and 28-40 days after the 3rd dose of vaccination. Neutralization antibody would also be detected to evaluate the seroprotection rates and antibody geometric mean concentrations. The safety of both immunization schedule will be monitored as well.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged 3 months old at the date of recruitment;
* with informed consent signed by parent(s) or guardians;
* parent(s) or guardians are able to attend all planned clinical appointments and obey and follow all study instructions;
* subjects have not been vaccinated with IPV vaccine, OPV vaccine, DTP vaccine and related vaccines;

Exclusion Criteria:

* subject who has a medical history with Hypersensitiveness, eclampsia, epilepsy, cerebropathia and neurological illness;
* allergic to any ingredient of vaccine or with allergy history to any vaccine;
* subjects with immunodeficency or suspected impairment of immunologic function (e.g. caused by HIV), or subjects are in the process of immunosuppressor therapy(Taking orally injecting of steroid hormone);
* administration of immunoglobulins within 30 days prior to this study;
* acute febrile disease(temperature ≥ 37.0°C) or infectious disease;
* have a clearly diagnosed history of thrombocytopenia or other coagulopathy, may cause contraindications for subcutaneous injection;
* any serious chronic illness, acute infectious diseases, or respiratory diseases;
* severe cardiovascular disease, liver and kidney diseases or diabetes mellitus with complications;
* any kind of infectious, purulent, or allergic skin diseases;
* any other factor that makes the investigator determines the subject is unsuitable for this study.

Ages: 3 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 702 (Estimated)
Dates: Start 2019-08-10 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate I | 1 month after the 3rd dose
  determine the rate of positive seroconversion against poliovirus type I, II and III of the 3 groups
Seroconversion rate II | 1 month after the 3rd dose
  determine the positive seroconversion rate of anti-pertussis toxoid , anti- filamentous hemagglutinin, anti-diphtheria toxoid and anti-tetanic antibody of the 3 groups
Neutralizing antibody titers I | 1 month after the 3rd dose
  Measure neutralizing antibody titers against poliovirus type I, II and III
Neutralizing antibody titers II | 1 month after the 3rd dose
  Measure neutralizing antibody titers against diphtheria, pertussis toxoid, pertussis filamentous hemagglutinin, and tetanic of the 3 groups

SECONDARY OUTCOMES:
safety outcomes | 6 months
  Adverse event following vaccinations

CONTACTS AND LOCATIONS:
Overall Officials: Shaobai ZHANG, Principal Investigator — Shaanxi Provincial Center for Disease Control and Prevention
Locations (1):
- Shaanxi Provincial Center for Disease Control and Prevention, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Liu X, Han S, Chen X, Sun L, Wang R, Shi X, Guo Y, Wang H, Chen H, Chang S, Xu X, Zhang C, Wang Y, Zhang D, Hu W, Zhang S. Immunogenicity and safety of co-administration with the Sabin-strain-based inactivated poliovirus vaccine (vero cell) and the diphtheria-tetanus-acellular pertussis vaccine in eligible children in China: a randomized, controlled, multicenter, non-inferiority trial. Front Immunol. 2025 Sep 3;16:1633170. doi: 10.3389/fimmu.2025.1633170. eCollection 2025. PMID 40969746